CLINICAL TRIAL: NCT00602667
Title: Risk-Adapted Therapy for Young Children With Embryonal Brain Tumors, Choroid Plexus Carcinoma, High Grade Glioma or Ependymoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Florida (Other); National Cancer Institute (NCI) (NIH); The Pew Charitable Trusts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJYC07; R01CA154619 (NIH); NCI-2011-01193 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2008-01-10; First posted 2008-01-28 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood pineoblastoma; childhood atypical teratoid/rhabdoid tumor; childhood choroid plexus tumor; childhood high grade glioma; newly diagnosed childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Rhabdoid Tumor; Choroid Plexus Neoplasms | interventions — Induction Chemotherapy; Methotrexate; Vincristine; Cisplatin; Cyclophosphamide; Carboplatin; Etoposide; Topotecan; Erlotinib Hydrochloride; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-Risk Patients (Experimental): Patients with GTR/M0 medulloblastoma, nodular desmoplastic or high grade glioma histology will receive induction chemotherapy and low-risk therapy.
  Note: Accrual to the low-risk medulloblastoma cohort is closed as of 12/2/2015. Accrual to the low-risk high grade glioma remains open.
  Interventions: Drug: Induction Chemotherapy; Drug: Low-Risk Therapy
- High-Risk Patients (Experimental): Patients with CNS metastatic disease will receive induction chemotherapy and high-risk therapy.
  Interventions: Drug: Induction Chemotherapy; Drug: High-Risk Therapy
- Intermediate-Risk Therapy (Experimental): Patients with M0 medulloblastoma or nodular desmoplastic histology with less than a GTR, other histologic diagnoses with no metastatic disease, will receive induction chemotherapy and intermediate-risk therapy.
  Interventions: Drug: Induction Chemotherapy; Drug: Intermediate-Risk Therapy

INTERVENTIONS:
Drug: Induction Chemotherapy — All patients will receive 4 identical cycles of induction chemotherapy including highdose (5 g/m2 or 2.5g/m2 for patients less than or equal to 31 days of age at enrollment) intravenous methotrexate and standard dose vincristine, cisplatin, and cyclophosphamide.
  Other Names: MTX (methotrexate); Oncovin(R) (vincristine); Platinol-AQ(R) (cisplatin); Cytoxan(R) (cyclophosphamide)
Drug: Low-Risk Therapy — Induction will be followed by further conventional chemotherapy with carboplatin, cyclophosphamide, and etoposide. After consolidation, patients will receive 6 cycles of oral maintenance chemotherapy with cyclophosphamide, topotecan, and depending on the diagnosis, either erlotinib or etoposide (VP-16).
  Other Names: Cytoxan(R) (cyclophosphamide); Paraplatin(R) (carboplatin); Vepesid(R), VP-16 (etoposide); Hycamptin(R) (topotecan); Tarceva(TM) (erlotinib)
  Arms: Low-Risk Patients
Drug: High-Risk Therapy — High risk patients will also receive vinblastine with each course of induction chemotherapy. Induction will be followed by either chemotherapy with targeted intravenous topotecan and cyclophosphamide or optional craniospinal irradiation (CSI). CSI will be offered only to patients who reach 3 years of age by the end of induction only. After consolidation, all patients will receive 6 cycles of oral maintenance chemotherapy with cyclophosphamide, topotecan, and depending on the diagnosis, either erlotinib or etoposide (VP-16).
  Other Names: Velban(R) (vinblastine); Cytoxan(R) (cyclophosphamide); Hycamptin(R) (topotecan); Tarceva(TM) (erlotinib); Vepesid(R), VP-16 (etoposide)
  Arms: High-Risk Patients
Drug: Intermediate-Risk Therapy — Induction will be followed by consolidation focal radiotherapy (RT) to the tumor bed. Patients less than 12 months old upon completion of induction will receive low risk chemotherapy to delay RT until the age of 12 months. After consolidation, patients will receive 6 cycles of oral maintenance chemotherapy with cyclophosphamide, topotecan, and depending on the diagnosis, either erlotinib or etoposide (VP-16).
  Note: The option to receive focal proton beam irradiation was suspended 10/29/2015. Focal photon beam irradiation continues as part of the treatment plan.
  Other Names: Cytoxan(R) (cyclophosphamide); Hycamptin(R) (topotecan); Tarceva(TM) (erlotinib); Vepesid(R), VP-16 (etoposide)
  Arms: Intermediate-Risk Therapy

SUMMARY:
RATIONALE: In this study a combination of anti-cancer drugs (chemotherapy) is used to treat brain tumors in young children. Using chemotherapy gives the brain more time to develop before radiation is given. The chemotherapy in this study includes the drug methotrexate. This drug was an important part of the two clinical trials which resulted in the best survival results for children less than 3 years of age with medulloblastoma. Most patients treated on this trial will also receive radiation which is carefully targeted to the area of the tumor. This type of radiation (focal conformal or proton beam radiotherapy) may result in fewer problems with thinking and learning than radiation to the whole brain and spinal cord.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy together with radiation therapy works in treating young patients with newly diagnosed central nervous system tumors.

DETAILED DESCRIPTION:
All patients with medulloblastoma who were diagnosed prior to their 3rd birthday will contribute to both the biology and therapeutic primary objectives of this protocol. Furthermore patients who were ≥3 and <5 years old at the time of diagnosis will also be included in the cohort for these primary objectives as long as they meet the eligibility criteria as outlined in Amendment 8.0 of this protocol. Patients in the 3-5 year old age cohort who enrolled on previous versions of this protocol and who do not meet the criteria as outlined in Amendment 8.0 of this protocol will be excluded from the outcome analyses of the biology and therapeutic primary objectives of the protocol.

OBJECTIVES:

Primary

* To identify patterns of methylation profiling that are associated with progression-free survival among young pediatric patients with medulloblastoma treated with risk-adapted therapy.
* To estimate the event-free survival distribution of young medulloblastoma patients treated with risk-adapted therapy.

Secondary

* To perform high-resolution genome-wide analyses of chromosomal abnormalities and gene expression patterns, and evaluate the relationship of these to other clinicopathological variables.
* To evaluate specific tumor types for molecular abnormalities with suspected prognostic or therapeutic significance.
* To evaluate the feasibility of collecting frozen and fixed tumor samples for analysis using high-resolution molecular biology tools.
* To estimate the event-free and overall survival of patients treated with the proposed risk-adapted therapy regimen, and to descriptively compare these survival rates to historical controls.
* To estimate the rates of local and distant disease progression in patients treated with focal radiotherapy (RT) to the post-operative tumor bed using a 5 mm clinical target volume margin.
* To estimate the objective response rate (sustained for 8 weeks) to induction chemotherapy including high-dose intravenous methotrexate for patients with residual or metastatic disease.
* To evaluate the feasibility and toxicity of administering low-dose intravenous vinblastine in conjunction with induction chemotherapy to patients with metastatic disease.
* To evaluate the feasibility and toxicity of administering consolidation therapy including cyclophosphamide and pharmacokinetically targeted topotecan to patients with metastatic disease, and to estimate the sustained (for 8 weeks) objective response rate (complete response and partial response) to such therapy in patients with measurable residual disease after induction.
* To evaluate the feasibility and toxicity of administering oral maintenance therapy in young children.
* To use quantitative magnetic resonance (MR) measures (volumetric, diffusion, and perfusion) of young brain tumor patients receiving chemotherapy including high-dose intravenous methotrexate to assess impact of treatment on developing brain.
* To investigate the feasibility of using PET as an in-vivo dosimetric and distal edge verification system for patients treated with proton beam therapy (for participants enrolled at St Jude only).

OUTLINE: This is a multicenter study. Patients are stratified according to disease risk (low-risk vs intermediate-risk vs high-risk). Therapy consists of risk adapted induction, consolidation and maintenance chemotherapy. Focal irradiation is given to intermediate risk patients who have reached at least 12 months of age upon completion of induction. Intermediate risk patients who have not will receive low risk chemotherapy to delay RT until the age of 12 months.

Patients may consent to provide tumor tissue and blood samples for biological studies. Tumor tissues are analyzed for the activation of the wnt signaling pathway (β-catenin), activation of the shh signaling pathway (Gli-1/SFRP1), and ERBB2; validation of novel patterns of gene expression via immunohistochemical (IHC) analysis; loss of chromosomes 6, 8p, 9q22, isochromosome 17q; amplification of MYCC, MYCN, and MYCL; validation of genetic abnormalities via interphase fluorescence in situ hybridization (iFISH); construction of gene expression profiles via microarray analysis; single nucleotide polymorphism (SNP) analysis for DNA purity and integrity using UV spectrophotometry and agarose gel electrophoresis; amplification of DNA via PCR and a combination of previously published and 'in-house' generated primers; potential oncogenes and tumor suppressor genes via DNA sequence analysis; expression of a number of cell signal proteins implicated in the biology of medulloblastoma via western blot; expression of additional proteins encoded by genes associated through SNP and gene expression array analysis with clinical disease behavior; and differential expression pattern of genes detected using microarray analysis via RT-PCR. DNA extraction and construction of tissue microarrays (TMAs) from tumor tissue will also be used for future IHC and FISH analysis. Blood samples are analyzed for constitutional DNA from patients whose tumors contain gene mutations via sequence analysis of constitutional DNA; cyclophosphamide and its metabolites via liquid chromatography mass spectroscopy method; topotecan lactone via isocratic high-performance liquid chromatography assay with fluorescence detection; and alpha-1-acid glycoprotein (AAGP) concentrations via immunoturbidimetric assay.

After completion of study treatment, patients are followed every 6 months for 5 years.

ELIGIBILITY:
Histologically confirmed newly diagnosed CNS tumors of any of the following :

* Medulloblastoma (all histologic subtypes, including medullomyoblastoma and melanotic medulloblastoma)
* Supratentorial primitive neuroectodermal tumor (PNET) (including CNS neuroblastoma or ganglioneuroblastoma, medulloepithelioma, and ependymoblastoma)
* Pineoblastoma
* Atypical teratoid rhabdoid tumor (ATRT)
* Choroid plexus carcinoma
* High grade glioma (including anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic ganglioglioma, pleomorphic xanthoastrocytoma with anaplastic features, high-grade astroblastoma , anaplastic pilocytic astrocytoma, malignant glioneuronal tumor, glioblastoma multiforme), or gliosarcoma,
* Ependymoma (including all ependymoma histological variants)
* Age < 3 years at time of diagnosis for all histological diagnosis. Medulloblastoma patients ≥ 3 and < 5years old at diagnosis who have non-metastatic disease with no more than 1cm2 of residual tumor are also eligible.

  * Meets criteria for 1 of the following risk groups:
* Low-risk group:

  * Histologically confirmed nodular desmoplastic medulloblastoma, including medulloblastoma with extensive nodularity

    * Focal areas of anaplasia or other atypical features suggesting more aggressive phenotype in a tumor otherwise considered nodular desmoplastic should be treated on the intermediate-risk group, with final risk stratification at the discretion of principal investigator and study pathologist
  * No evidence of CNS metastasis 7 to 28 days after surgery by MRI and cytologic examination of lumbar cerebrospinal fluid (CSF)

    * Ventricular CSF from a shunt or Ommaya reservoir may be used to rule out M1 disease when lumbar puncture is medically contraindicated
    * Intermediate-risk group assignment when there is no other evidence of metastasis and CSF sampling is not possible
  * Gross total resection, defined as residual tumor or imaging abnormality (not definitive for residual tumor) with a size of < 1 cm2 confirmed on postoperative CT scan or MRI
  * Brain stem invasion by the tumor in the absence of imaging evidence of residual tumor (tumor size < 1 cm2) and otherwise meets criteria for the low-risk group, the patient will be classified as low-risk
  * Desmoplastic medulloblastoma patients who are ≥3 -<5 years of age will NOT be eligible for the low risk arm of the protocol.
* Intermediate-risk group:

  * Histologically confirmed nodular desmoplastic medulloblastoma with less than gross total resection and no evidence of metastasis
  * Any eligible histologic diagnosis other than desmoplastic medulloblastoma with no evidence of CNS metastasis
  * Medulloblastoma patients who are ≥3 and < 5 yrs of age irrespective of histology and with no evidence of CNS metastasis
* High-risk group:

  * Any eligible histologic diagnosis with evidence of CNS metastasis
  * Patients with extraneural metastasis are eligible for treatment on the high-risk group

PATIENT CHARACTERISTICS:

* Lansky performance status ≥ 30 (except for posterior fossa syndrome)
* WBC > 2,000/mm3
* Platelets > 50,000/mm3 (without support)
* Hemoglobin > 8 g/dL (with or without support)
* ANC > 500/mm3
* Serum creatinine < 3 times upper limit of normal (ULN)
* ALT < 5 times ULN
* Total bilirubin < 3 times ULN

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 31 days since prior definitive surgery
* No prior radiotherapy or chemotherapy other than corticosteroid therapy

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, MD, Study Chair — St. Jude Children's Research Hospital
Locations (6):
- United States (5):
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospitals and Clinics of Minnesota - St. Paul, Saint Paul, Minnesota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
- Lady Cilento Children's Hospital, Brisbane, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Ali JS, Ashford JM, Swain MA, Harder LL, Carlson-Green BL, Miller JM, Wallace J, Kaner RJ, Billups CA, Onar-Thomas A, Merchant TE, Gajjar A, Conklin HM. Predictors of Cognitive Performance Among Infants Treated for Brain Tumors: Findings From a Multisite, Prospective, Longitudinal Trial. J Clin Oncol. 2021 Jul 20;39(21):2350-2358. doi: 10.1200/JCO.20.01687. Epub 2021 May 4. PMID 33945291
- [Derived] Kumar R, Smith KS, Deng M, Terhune C, Robinson GW, Orr BA, Liu APY, Lin T, Billups CA, Chintagumpala M, Bowers DC, Hassall TE, Hansford JR, Khuong-Quang DA, Crawford JR, Bendel AE, Gururangan S, Schroeder K, Bouffet E, Bartels U, Fisher MJ, Cohn R, Partap S, Kellie SJ, McCowage G, Paulino AC, Rutkowski S, Fleischhack G, Dhall G, Klesse LJ, Leary S, Nazarian J, Kool M, Wesseling P, Ryzhova M, Zheludkova O, Golanov AV, McLendon RE, Packer RJ, Dunham C, Hukin J, Fouladi M, Faria CC, Pimentel J, Walter AW, Jabado N, Cho YJ, Perreault S, Croul SE, Zapotocky M, Hawkins C, Tabori U, Taylor MD, Pfister SM, Klimo P Jr, Boop FA, Ellison DW, Merchant TE, Onar-Thomas A, Korshunov A, Jones DTW, Gajjar A, Ramaswamy V, Northcott PA. Clinical Outcomes and Patient-Matched Molecular Composition of Relapsed Medulloblastoma. J Clin Oncol. 2021 Mar 1;39(7):807-821. doi: 10.1200/JCO.20.01359. Epub 2021 Jan 27. PMID 33502920
- [Derived] Robinson GW, Rudneva VA, Buchhalter I, Billups CA, Waszak SM, Smith KS, Bowers DC, Bendel A, Fisher PG, Partap S, Crawford JR, Hassall T, Indelicato DJ, Boop F, Klimo P, Sabin ND, Patay Z, Merchant TE, Stewart CF, Orr BA, Korbel JO, Jones DTW, Sharma T, Lichter P, Kool M, Korshunov A, Pfister SM, Gilbertson RJ, Sanders RP, Onar-Thomas A, Ellison DW, Gajjar A, Northcott PA. Risk-adapted therapy for young children with medulloblastoma (SJYC07): therapeutic and molecular outcomes from a multicentre, phase 2 trial. Lancet Oncol. 2018 Jun;19(6):768-784. doi: 10.1016/S1470-2045(18)30204-3. Epub 2018 May 16. PMID 29778738
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 293 participants were enrolled between December 17, 2007 and April 19, 2017.
Pre-assignment Details: Of the 293 participants enrolled, 3 were ineligible and removed from study, leaving 290 eligible patients. Eighty-one (81) of the 290 eligible patients enrolled had histologically confirmed medulloblastoma; medulloblastoma patients are the focus of the primary study objectives.
Groups:
- Low-Risk Group: Patients with gross total resection (GTR)/no evidence of metastatic (M0) medulloblastoma, nodular desmoplastic or high grade glioma histology will receive induction chemotherapy and low-risk therapy.
- Intermediate-Risk Group: Patients with M0 medulloblastoma or nodular desmoplastic histology with less than a GTR, other histologic diagnoses with no metastatic disease, will receive induction chemotherapy and intermediate-risk therapy.
- High-Risk Group: Patients with central nervous system (CNS) metastatic disease will receive induction chemotherapy and high-risk therapy.
Period: Overall Study
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Started | 57 | 156 | 77
Completed | 38 | 75 | 14
Not Completed | 19 | 81 | 63
Not completed — Still on Therapy | 0 | 2 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Family request | 3 | 25 | 6
Not completed — Excessive toxicity | 1 | 1 | 0
Not completed — Second malignancy | 0 | 1 | 0
Not completed — Physician Decision | 2 | 3 | 8
Not completed — Progressive disease | 13 | 48 | 45
Not completed — Progressive disease prior to therapy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were patients with newly diagnosed tumors of the CNS, including medulloblastoma, supratentorial primitive neuroectodermal tumor (PNET), pineoblastoma, atypical teratoid rhabdoid tumor (ATRT), choroid plexus carcinoma, ependymoma, and high-grade glioma. All eligible patients enrolled were included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group | Total
Number analyzed (Participants) | 57 | 156 | 77 | 290
Age, Continuous [Mean (Standard Deviation); unit: months] | 17.0 (10.0) | 22.9 (12.8) | 19.3 (10.4) | 20.8 (11.9)
Age, Continuous [Median (Full Range); unit: months] | 16.1 [0.2 to 35.2] | 21.9 [1.8 to 60.6] | 20.0 [0.9 to 36.9] | 20.1 [0.2 to 60.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 66 | 43 | 131
  Male | 35 | 90 | 34 | 159
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Mexican/Chicano | 0 | 5 | 2 | 7
  Ethnicity: NOS Spanish, Hispanic, Latino | 7 | 16 | 7 | 30
  Ethnicity: Non Spanish speaking, Non Hispanic | 47 | 120 | 64 | 231
  Ethnicity: Puerto Rican | 1 | 2 | 1 | 4
  Ethnicity: South or Central American | 0 | 2 | 0 | 2
  Ethnicity: Unknown | 2 | 11 | 3 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaskan/White | 1 | 0 | 0 | 1
  Race: American Indian/Alaskan Native | 0 | 1 | 0 | 1
  Race: Asian | 3 | 6 | 1 | 10
  Race: Asian and White | 0 | 2 | 2 | 4
  Race: Black | 6 | 14 | 10 | 30
  Race: Black and White | 0 | 1 | 0 | 1
  Race: Multiple Race (NOS) | 1 | 7 | 1 | 9
  Race: Other | 2 | 4 | 1 | 7
  Race: Pacific Islander | 1 | 0 | 0 | 1
  Race: Unknown | 2 | 3 | 1 | 6
  Race: White | 41 | 118 | 61 | 220

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability of Progression-free Survival (PFS) for Medulloblastoma Patients
Description: Progression was defined as 25% increase in the size of any measurable lesion; the appearance of a new lesion; or the conversion of negative cerebrospinal fluid (CSF) cytology to positive. Defined as the time interval from date on treatment until the date of first progression, medulloblastoma-related death or date of last contact for patients who have not experienced an event. All eligible medulloblastoma patients who received any methotrexate are included in this analysis.
Time Frame: From date on treatment until date of first progression or relapse or disease related death or date of last contact, estimated at 1 year after treatment
Population: All eligible medulloblastoma patients started methotrexate and were included (n=81). PFS estimates are reported by risk group.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Groups:
- Low-Risk Group: Medulloblastoma patients <3 years of age; histological diagnosis of desmoplastic nodular (DN)/medulloblastoma with extensive nodularity (MBEN); no evidence of metastatic disease (M0); and a surgical gross total resection (GTR) or near total resection (NTR) defined as residual tumor or imaging abnormality (not definite for residual tumor) with a size of less than 1 cm^2 on post-op computed tomography (CT) or magnetic resonance imaging (MRI) [R0])
- Intermediate-Risk Group: Medulloblastoma patients <3 years of age, M0, and either R0 resection with any other medullo histology other than DN/MBEN (i.e., classic or large cell anaplastic (LCA)), or with a subtotal resection (with a residual tumor or imaging abnormality with a size of >1 cm^2 on post-op imaging (R+), and DN/MBEN). Children 3-5 years of age were also included in this group High Risk
- High-Risk Group: Medulloblastoma patients <3 years of age with evidence of metastatic disease
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 23 | 32 | 26
Percent Probability | 73.9 [56.5 to 91.3] | 46.9 [30.2 to 63.6] | 30.8 [14.1 to 47.5]

2. Primary Outcome: Percent Probability of Progression-free Survival (PFS) for Medulloblastoma Patients by DNA Methylation Subgroup
Description: Defined as the time interval from date on treatment until the date of first progression, medulloblastoma-related death or date of last contact for patients who have not experienced an event. Eligible medulloblastoma patients who received any methotrexate and had molecularly confirmed medulloblastoma are included in this analysis. Five patients were excluded as 3 had no archival tissue available and 2 were found to not be medulloblastoma by methylation profile.
Time Frame: From date on treatment to date of first progression or relapse or disease related death or date of last contact, estimated at 1 year after treatment
Population: Eligible patients with molecularly confirmed medulloblastoma (n=76) were included. PFS estimates are reported by methylation subgroup and risk group. There were no low-risk group 3 or group 4 patients.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Groups:
- Low-risk SHH Patients: Sonic hedgehog (SHH) medulloblastoma subgroup patients in the low-risk group
- Intermediate-risk SHH Patients: Sonic hedgehog (SHH) medulloblastoma subgroup patients in the intermediate-risk group
- High-risk SHH Patients: Sonic hedgehog (SHH) medulloblastoma subgroup patients in the high-risk group
- Low-risk Group 3 Patients: Group 3 (G3) medulloblastoma subgroup patients in the low-risk group
- Intermediate-risk Group 3 Patients: Group 3 medulloblastoma subgroup patients in the intermediate-risk group
- High-risk Group 3 Patients: Group 3 medulloblastoma subgroup patients in the high-risk group
- Low-risk Group 4 Patients: Group 4 (G4) medulloblastoma subgroup patients in the low-risk group
- Intermediate-risk Group 4 Patients: Group 4 (G4) medulloblastoma subgroup patients in the intermediate-risk group
- High-risk Group 4 Patients: Group 4 medulloblastoma subgroup patients in the high-risk group
Arm/Group | Low-risk SHH Patients | Intermediate-risk SHH Patients | High-risk SHH Patients | Low-risk Group 3 Patients | Intermediate-risk Group 3 Patients | High-risk Group 3 Patients | Low-risk Group 4 Patients | Intermediate-risk Group 4 Patients | High-risk Group 4 Patients
Number analyzed (Participants) | 23 | 8 | 11 | 0 | 13 | 11 | 0 | 8 | 2
Percent Probability | 73.9 [56.5 to 91.3] | 50.0 [19.0 to 81.0] | 54.5 [27.3 to 81.7] |  | 30.8 [8.5 to 53.1] | 9.1 [0.0 to 21.1] |  | 62.5 [31.9 to 93.1] | 50.0 [1.0 to 99.0]

3. Primary Outcome: Percent Probability of Event-free Survival (EFS) for Medulloblastoma Patients
Description: Defined as the time interval from date on treatment until the date of first progression, second malignancy or death due to any cause; or date of last contact for patients who have not experienced an event. All eligible medulloblastoma patients who received any methotrexate are included in this analysis.
Time Frame: From date on treatment to date of first progression, relapse, second malignancy or death from any cause or to date of last contact, estimated at 1 year after
Population: Eligible medulloblastoma patients (n=81) were included. EFS estimates are reported by risk group.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 23 | 32 | 26
Percent Probability | 73.9 [56.5 to 91.3] | 46.9 [30.2 to 63.6] | 30.8 [14.1 to 47.5]

4. Secondary Outcome: Number of Participants With Chromosomal Abnormalities
Description: Amplifications and deletions (gains and losses) for chromosomes of interest are shown in the table of measured values.
Time Frame: Based on samples obtained at the time of initial surgery or repeat surgery prior to treatment
Population: Eligible medulloblastoma patients (n=81) were included in these analyses. 23 of 23 low risk patients had data available for this objective, as did 27/32 and 24/26 intermediate and high risk patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 23 | 32 | 26
Participants
  chr2p gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr2p gain/amplification | 5 | 1 | 6
  chr2p loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr2p loss/deletion | 0 | 2 | 0
  chr2q gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr2q gain/amplification | 5 | 1 | 6
  chr2q loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr2q loss/deletion | 0 | 2 | 0
  chr6p gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr6p gain/amplification | 1 | 3 | 3
  chr6p loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr6p loss/deletion | 0 | 0 | 2
  chr6q gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr6q gain/amplification | 1 | 3 | 3
  chr6q loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr6q loss/deletion | 0 | 0 | 2
  chr8p gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr8p gain/amplification | 1 | 2 | 0
  chr8p loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr8p loss/deletion | 0 | 6 | 8
  chr8q gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr8q gain/amplification | 1 | 3 | 0
  chr8q loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr8q loss/deletion | 0 | 5 | 7
  chr9p gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr9p gain/amplification | 4 | 6 | 3
  chr9p loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr9p loss/deletion | 4 | 0 | 3
  chr9q gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr9q gain/amplification | 2 | 1 | 1
  chr9q loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr9q loss/deletion | 6 | 5 | 5
  chr10p gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr10p gain/amplification | 0 | 0 | 0
  chr10p loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr10p loss/deletion | 0 | 5 | 7
  chr10q gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr10q gain/amplification | 0 | 0 | 0
  chr10q loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr10q loss/deletion | 3 | 7 | 9
  chr20p gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr20p gain/amplification | 0 | 0 | 0
  chr20p loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr20p loss/deletion | 2 | 4 | 5
  chr20q gain/amplification: number analyzed (Participants) | 23 | 27 | 24
  chr20q gain/amplification | 0 | 0 | 0
  chr20q loss/deletion: number analyzed (Participants) | 23 | 27 | 24
  chr20q loss/deletion | 1 | 3 | 5

5. Secondary Outcome: Numbers of Patients With Gene Alterations
Description: Gene alterations, which include single nucleotide variants (SNPs), amplifications, deletions, translocations, indels, and germline alterations are shown for specific genes of interest in the results table.
Time Frame: Based on samples obtained at the time of initial surgery or repeat surgery prior to treatment
Population: Eligible medulloblastoma patients (n=81) were included in these analyses. Not all patients had data available for each gene.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 23 | 32 | 26
Participants
  PTCH1 alteration: number analyzed (Participants) | 23 | 28 | 24
  PTCH1 alteration | 7 | 4 | 3
  SUFU alteration: number analyzed (Participants) | 23 | 28 | 24
  SUFU alteration | 6 | 1 | 1
  KMT2D alteration: number analyzed (Participants) | 22 | 20 | 17
  KMT2D alteration | 5 | 1 | 3
  SMO alteration: number analyzed (Participants) | 22 | 20 | 17
  SMO alteration | 2 | 0 | 1
  BCOR alteration: number analyzed (Participants) | 22 | 20 | 17
  BCOR alteration | 1 | 0 | 0
  PTEN alteration: number analyzed (Participants) | 23 | 28 | 24
  PTEN alteration | 1 | 0 | 0
  BRCA2 alteration: number analyzed (Participants) | 22 | 20 | 17
  BRCA2 alteration | 0 | 0 | 0
  GLI2 alteration: number analyzed (Participants) | 23 | 26 | 23
  GLI2 alteration | 0 | 0 | 0
  SMARCA4 alteration: number analyzed (Participants) | 22 | 20 | 17
  SMARCA4 alteration | 2 | 1 | 0
  TP53 alteration: number analyzed (Participants) | 23 | 28 | 24
  TP53 alteration | 0 | 0 | 0
  MYCN alteration: number analyzed (Participants) | 23 | 28 | 24
  MYCN alteration | 0 | 1 | 1

6. Secondary Outcome: Numbers of Patients With Molecular Abnormalities by Tumor Type
Description: Alterations included single nucleotide variants (SNPs), amplifications, deletions, translocations, indels, and germline alterations. Cytogenetic information shows gains and losses as specified in the table of measured values.
Time Frame: Based on samples obtained at the time of initial surgery or repeat surgery prior to treatment
Population: Eligible patients with molecularly confirmed medulloblastoma (n=76) were included in these analyses. Not all patients had data available for each gene.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-risk SHH Patients | Intermediate-risk SHH Patients | High-risk SHH Patients | Low-risk Group 3 Patients | Intermediate-risk Group 3 Patients | High-risk Group 3 Patients | Low-risk Group 4 Patients | Intermediate-risk Group 4 Patients | High-risk Group 4 Patients
Number analyzed (Participants) | 23 | 8 | 11 | 0 | 13 | 11 | 0 | 8 | 2
Participants
  PTCH1 alteration: number analyzed (Participants) | 23 | 8 | 11 | 0 | 12 | 11 | 0 | 8 | 2
  PTCH1 alteration | 7 | 4 | 3 |  | 0 | 0 |  | 0 | 0
  SUFU alteration: number analyzed (Participants) | 23 | 8 | 11 | 0 | 12 | 11 | 0 | 8 | 2
  SUFU alteration | 6 | 1 | 1 |  | 0 | 0 |  | 0 | 0
  KMT2D alteration: number analyzed (Participants) | 22 | 6 | 10 | 0 | 9 | 6 | 0 | 5 | 2
  KMT2D alteration | 5 | 1 | 3 |  | 0 | 0 |  | 0 | 0
  SMO alteration: number analyzed (Participants) | 22 | 6 | 10 | 0 | 9 | 6 | 0 | 5 | 1
  SMO alteration | 2 | 0 | 1 |  | 0 | 0 |  | 0 | 0
  BCOR alteration: number analyzed (Participants) | 22 | 6 | 10 | 0 | 9 | 6 | 0 | 5 | 1
  BCOR alteration | 1 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  PTEN alteration: number analyzed (Participants) | 23 | 8 | 11 | 0 | 12 | 11 | 0 | 8 | 2
  PTEN alteration | 1 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  BRCA2 alteration: number analyzed (Participants) | 22 | 6 | 10 | 0 | 9 | 6 | 0 | 5 | 1
  BRCA2 alteration | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  GLI2 alteration: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  GLI2 alteration | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  SMARCA4 alteration: number analyzed (Participants) | 22 | 6 | 10 | 0 | 9 | 6 | 0 | 5 | 1
  SMARCA4 alteration | 2 | 0 | 0 |  | 1 | 0 |  | 0 | 0
  TP53 alteration: number analyzed (Participants) | 23 | 8 | 11 | 0 | 12 | 11 | 0 | 8 | 2
  TP53 alteration | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  MYCN amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 12 | 11 | 0 | 8 | 2
  MYCN amplification | 0 | 1 | 0 |  | 0 | 1 |  | 0 | 0
  chr2p gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr2p gain/amplification | 5 | 0 | 4 |  | 0 | 1 |  | 0 | 0
  chr2p loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr2p loss/deletion | 0 | 0 | 0 |  | 1 | 0 |  | 1 | 0
  chr2q gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr2q gain/amplification | 5 | 0 | 4 |  | 0 | 1 |  | 0 | 0
  chr2q loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr2q loss/deletion | 0 | 0 | 0 |  | 1 | 0 |  | 1 | 0
  chr6p gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr6p gain/amplification | 1 | 0 | 0 |  | 2 | 3 |  | 1 | 0
  chr6p loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr6p loss/deletion | 0 | 0 | 0 |  | 0 | 2 |  | 0 | 0
  chr6q gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr6q gain/amplification | 1 | 0 | 0 |  | 2 | 3 |  | 1 | 0
  chr6q loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr6q loss/deletion | 0 | 0 | 0 |  | 0 | 2 |  | 0 | 0
  chr8p gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr8p gain/amplification | 1 | 0 | 0 |  | 1 | 0 |  | 0 | 0
  chr8p loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr8p loss/deletion | 0 | 0 | 0 |  | 2 | 7 |  | 4 | 1
  chr8q gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr8q gain/amplification | 1 | 0 | 0 |  | 2 | 0 |  | 0 | 0
  chr8q loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr8q loss/deletion | 0 | 0 | 0 |  | 1 | 6 |  | 4 | 1
  chr9p gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr9p gain/amplification | 4 | 4 | 3 |  | 1 | 0 |  | 1 | 0
  chr9p loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr9p loss/deletion | 4 | 0 | 0 |  | 0 | 3 |  | 0 | 0
  chr9q gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr9q gain/amplification | 2 | 0 | 1 |  | 0 | 0 |  | 1 | 0
  chr9q loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr9q loss/deletion | 6 | 5 | 2 |  | 0 | 3 |  | 0 | 0
  chr10p gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr10p gain/amplification | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  chr10p loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr10p loss/deletion | 0 | 0 | 0 |  | 5 | 7 |  | 0 | 0
  chr10q gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr10q gain/amplification | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  chr10q loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr10q loss/deletion | 3 | 2 | 1 |  | 5 | 8 |  | 0 | 0
  chr20p gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr20p gain/amplification | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  chr20p loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr20p loss/deletion | 2 | 1 | 1 |  | 3 | 4 |  | 0 | 0
  chr20q gain/amplification: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr20q gain/amplification | 0 | 0 | 0 |  | 0 | 0 |  | 0 | 0
  chr20q loss/deletion: number analyzed (Participants) | 23 | 8 | 11 | 0 | 11 | 11 | 0 | 7 | 1
  chr20q loss/deletion | 1 | 0 | 1 |  | 3 | 4 |  | 0 | 0

7. Secondary Outcome: Number of Successful Collections for Frozen and Fixed Tumor Samples
Description: Successful collections will be defined as the number of patients who have frozen/fixed tumor samples available.
Time Frame: Based on samples obtained at the time of initial surgery or repeat surgery prior to treatment
Population: All eligible patients enrolled (n=290) were included in this analysis. The numbers of patients with pre-study samples were considered for these results.
Measure: Count of Participants; unit: Participants
Groups:
- Low-Risk Group: Patients with gross total resection (GTR)/no evidence of metastatic disease (M0) medulloblastoma, nodular desmoplastic or high grade glioma histology will receive induction chemotherapy and low-risk therapy.
- Intermediate-Risk Group: Patients with (M0) medulloblastoma or nodular desmoplastic histology with less than a GTR, other histologic diagnoses with no metastatic disease, will receive induction chemotherapy and intermediate-risk therapy.
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 57 | 156 | 77
Participants
  Number with frozen tumor tissue | 27 | 73 | 32
  Number with fixed tumor tissue | 54 | 153 | 71

8. Secondary Outcome: Event-free Survival (EFS) Compared to Historical Controls
Description: EFS was measured from the date of initial treatment to the earliest date of disease progression, second malignancy or death for patients who fail; and to the date of last contact for patients who remain at risk for failure. 1-year EFS estimates are reported by risk group. EFS was compared to St. Jude historical cohorts by risk group using hazard ratios with 95% confidence intervals.
Time Frame: From date on treatment until date of first event (progression, second malignancy or death) or until date of last contact, assessed up to 10 years
Population: Eligible medulloblastoma patients who received any methotrexate were included in this analysis. Hazard ratios with 95% confidence intervals are reported and compare SJYC07 patients to historical controls in each risk group. As there were too few low-risk historical controls, no hazard ratio is included for the low-risk group.
Measure: Number (95% Confidence Interval); unit: Percent probability
Groups:
- SJYC07 Low-risk Medulloblastoma Patients: Medulloblastoma patients <3 years of age; histological diagnosis of desmoplastic nodular (DN)/medulloblastoma with extensive nodularity (MBEN); no evidence of metastatic disease (M0); and a surgical gross total resection (GTR) or near total resection (NTR) defined as residual tumor or imaging abnormality (not definite for residual tumor) with a size of less than 1 cm^2 on post-op computed tomography (CT) or magnetic resonance imaging (MRI) [R0])
- SJYC07 Intermediate-risk Medulloblastoma Patients: SJYC07 medulloblastoma patients <3 years of age, no evidence of metastatic disease (M0), and either R0 resection with any other medullo histology other than histological diagnosis of desmoplastic nodular (DN)/medulloblastoma with extensive nodularity (MBEN) (i.e., classic or large cell anaplastic (LCA)), or with a subtotal resection (with a residual tumor or imaging abnormality with a size of >1 cm^2 on post-op imaging (R+), and DN/MBEN). Children 3-5 years of age were also included in this group
- SJYC07 High-risk Medulloblastoma Patients: SJYC07 medulloblastoma patients <3 years of age with evidence of metastatic disease
Arm/Group | SJYC07 Low-risk Medulloblastoma Patients | SJYC07 Intermediate-risk Medulloblastoma Patients | SJYC07 High-risk Medulloblastoma Patients
Number analyzed (Participants) | 23 | 32 | 26
Percent probability | 73.9 [56.5 to 91.3] | 46.9 [30.2 to 63.6] | 30.8 [14.1 to 47.5]
Statistical Analysis 1: Comparison: SJYC07 Intermediate-risk Medulloblastoma Patients; The historical control included 10 medulloblastoma patients treated during 1998-2006 who would have been classified as intermediate risk according to SJYC07 criteria (section 13.1.3 of protocol); Test type: Other; Hazard Ratio (HR) = 4.99, 95% CI 2-sided [1.17 to 21.23]
Statistical Analysis 2: Comparison: SJYC07 High-risk Medulloblastoma Patients; The historical control included 14 medulloblastoma patients treated during 1998-2006 who would have been classified as high risk according to SJYC07 criteria (section 13.1.3 of protocol); Test type: Other; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.40 to 1.84]

9. Secondary Outcome: Overall Survival (OS) Compared to Historical Controls
Description: OS was measured from the date of initial treatment to date of death or to date of last contact for survivors. 1-year OS estimates were reported by risk group. OS was compared to St. Jude historical cohorts by risk group using hazard ratios with 95% confidence intervals.
Time Frame: 1 year after treatment initiation of last patient
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | SJYC07 Low-risk Medulloblastoma Patients | SJYC07 Intermediate-risk Medulloblastoma Patients | SJYC07 High-risk Medulloblastoma Patients
Number analyzed (Participants) | 23 | 32 | 26
Percent probability | 100 [100 to 100] | 84.4 [72.1 to 96.7] | 61.5 [43.9 to 79.1]
Statistical Analysis 1: Comparison: SJYC07 Intermediate-risk Medulloblastoma Patients; [analysis description as in outcome 8, analysis 1]; Test type: Other; Hazard Ratio (HR) = 1.85, 95% CI 2-sided [0.42 to 8.22]
Statistical Analysis 2: Comparison: SJYC07 High-risk Medulloblastoma Patients; [analysis description as in outcome 8, analysis 2]; Test type: Other; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.31 to 1.79]

10. Secondary Outcome: Percentage of Patients With Objective Responses Rate to Induction Chemotherapy
Description: For patients treated in the intermediate and high risk strata with residual or metastatic disease we will estimate the stratum-specific objective response rate (complete response (CR) or partial response [ PR]). All patients who receive at least 1 -dose of methotrexate are evaluable for response. Objective responses must be sustained for at least eight weeks.
Time Frame: From on-study date to 2 months after completion of induction chemotherapy (up to 4 months after on-study date)
Population: Eligible intermediate and high risk group patients who received at least 1 dose of methotrexate were included in this analysis. One of the high risk patients did not start therapy and was excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Intermediate-Risk Group: Patients with no evidence of metastatic disease (M0) medulloblastoma or nodular desmoplastic histology with less than a gross total resection (GTR), other histologic diagnoses with no metastatic disease
- High-Risk Group: Patients with central nervous system (CNS) metastatic disease
Arm/Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 156 | 76
Percentage of patients | 58.3 [50.2 to 66.2] | 21.1 [12.5 to 31.8]

11. Secondary Outcome: Feasibility and Toxicity of Administering Vinblastine With Induction Chemotherapy for Patients With Metastatic Disease as Measured by the Percentage of Courses Delayed for More Than 7 Days Due to Toxicity
Description: For the subset of patients with metastatic disease (high-risk group patients), during induction, the proportion percentage of courses during which subsequent chemotherapy administration was delayed for more than 7 days due to toxicity will be calculated. Patients were to receive 4 courses of induction and then consolidation chemotherapy.
Time Frame: From on-study date up to 4 months after on-study date
Population: Eligible high-risk group patients who started therapy were included in this analysis (n=76). 1 patient enrolled on the high-risk arm did not start therapy due to early disease progression and was excluded. Courses 2-4 of induction and the 1st consolidation course were used in this analysis. 76 patients (with 263 courses) were included.
Measure: Number (95% Confidence Interval); unit: Percentage of courses delayed
Units Other Than Participants: courses
Arm/Group | High-Risk Group
Number analyzed (Participants) | 76
Number analyzed (courses) | 263
Percentage of courses delayed | 3.8 [1.8 to 6.9]

12. Secondary Outcome: Feasibility and Toxicity of Administering Consolidation Therapy Including Cyclophosphamide and Pharmacokinetically Targeted Topotecan to Patients With Metastatic Disease Based on the Percentage of Courses Delayed for More Than 7 Days Due to Toxicity
Description: For the subset of patients with metastatic disease (high-risk group patients), during consolidation, we will calculate the number and proportion of courses during which subsequent chemotherapy administration was delayed for more than 7 days due to toxicity. Patients were to received 2 courses of consolidation chemotherapy and then maintenance therapy.
Time Frame: At completion of consolidation therapy (up to 6 months after on-study date)
Population: Eligible high-risk group patients who started therapy were included. Course 2 of consolidation and the 1st course of maintenance were used in this analysis and assessed for delays >7 days due to toxicity. Of the 76 high-risk patients that started induction therapy, 50 started consolidation (with 47 courses included in this analysis).
Measure: Number (95% Confidence Interval); unit: Percentage of courses delayed
Units Other Than Participants: courses
Arm/Group | High-Risk Group
Number analyzed (Participants) | 50
Number analyzed (courses) | 47
Percentage of courses delayed | 2.6 [0.5 to 8.5]

13. Secondary Outcome: Percent of Patients With Sustained Objective Responses Rate After Consolidation
Description: For patients enrolled on the high-risk arm with measurable residual disease after induction treated with consolidation therapy, we will estimate the objective response (complete response (CR)/partial response (PR)) rate after consolidation therapy with a 95% confidence interval. Objective responses must be sustained for at least eight weeks. All patients who receive at least 1 dose of cyclophosphamide or topotecan during consolidation are evaluable for response.
Time Frame: 8 weeks after completion of consolidation therapy (up to 8 months after on-study date)
Population: Of the 50 high-risk patients that started consolidation chemotherapy, 38 had measurable residual disease after induction and were included in this result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-Risk Group
Number analyzed (Participants) | 38
percentage of participants | 13.2 [4.4 to 28.1]

14. Secondary Outcome: Feasibility and Toxicity of Administering Oral Maintenance Therapy in Children <3 Years of Age as Measured by the Percentage of Total Scheduled Maintenance Doses Received
Description: These data are based on patient diaries. For children <3 years of age, we will calculate the percentage of total scheduled doses each patient received per course for each of the oral maintenance courses and report the overall average number percentage of doses received per course across patients. If patients received all planned doses, their percentage would be 100%. If the average percentage was less than 75%, then feasibility would be in question.
Time Frame: From start of oral maintenance therapy (approximately 6 months after on-study date) to completion of oral maintenance therapy (up to 1 year after on-study date)
Population: Eligible patients less than 3 years of age (n=273) constituted the study population for this analysis; 167 of these patients started the first course of maintenance and were included in this analysis (50 low-risk, 87 intermediate-risk, and 30 high-risk patients).
Measure: Mean (Standard Deviation); unit: Percentage of scheduled doses received
Groups:
- Low-Risk Group: Patients <3 years of age with gross total resection (GTR)/no evidence of metastatic disease (M0) medulloblastoma, nodular desmoplastic or high grade glioma histology will receive induction chemotherapy and low-risk therapy.
- Intermediate-Risk Group: Patients <3 years of age with M0 medulloblastoma or nodular desmoplastic histology with less than a GTR, other histologic diagnoses with no metastatic disease, will receive induction chemotherapy and intermediate-risk therapy.
- High-Risk Group: Patients <3 years of age with central nervous system (CNS) metastatic disease will receive induction chemotherapy and high-risk therapy
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 50 | 87 | 30
Percentage of scheduled doses received | 96 (8) | 91 (23) | 98 (4)

15. Secondary Outcome: Percent of PET Scans With Loss of Signal Intensity
Description: Measures will be analyzed for intermediate risk participants who receive proton beam therapy (PBT) and who consent. This objective aims to assess the feasibility of using post-proton beam therapy (PBT) positron emission tomography (PET) as an in-vivo dosimetric and distal edge verification system in this patient population. To quantify the decay in signal, 134 scans from 53 patients were analyzed by recording the mean activation value (MAV), the average recorded PET signal from activation, within the target volume. With each patient being given the same dose, the percent standard deviation in the MAV can serve as a quantitative representation of signal loss due to radioactive decay.
Time Frame: Up to 3 times during RT consolidation
Population: Intermediate risk patients treated at St. Jude were eligible to receive proton beam therapy through referral to the University of Florida Proton Therapy Institute. Patients electing to receive PBT and post-treatment PET scans after the delivery of one treatment beam were included in the analysis.
Measure: Mean (Standard Deviation); unit: mean activation value (MAV)
Units Other Than Participants: Scans
Groups:
- Intermediate Risk Group: Patients with M0 medulloblastoma or nodular desmoplastic histology with less than a GTR, other histologic diagnoses with no metastatic disease
Arm/Group | Intermediate Risk Group
Number analyzed (Participants) | 53
Number analyzed (Scans) | 134
mean activation value (MAV) | 60 (27)

16. Secondary Outcome: Concentration of Cerebrospinal Fluid Neurotransmitters
Description: Concentrations of various neurotransmitters in cerebrospinal fluid were measured at 5 timepoints. The median concentration of each neurotransmitter at each time point was calculated and provided with a full range.
Time Frame: Baseline, at the completion of therapy, and every 12 months up to 36 months after off therapy date
Population: Eligible patients who had cerebrospinal fluid neurotransmitter studies performed. Seventeen patients had studies performed.
Measure: Median (Full Range); unit: ng/ml
Groups:
- Patients With Neurotransmitter Studies: Patients with neurotransmitter studies
Arm/Group | Patients With Neurotransmitter Studies
Number analyzed (Participants) | 17
ng/ml
  Dopamine concentration at baseline: number analyzed (Participants) | 12
  Dopamine concentration at baseline | 3.16 [0.18 to 4586.18]
  Dopamine concentration at completion of treatment: number analyzed (Participants) | 12
  Dopamine concentration at completion of treatment | 3.70 [0.82 to 39.16]
  Dopamine concentration at 12 months off treatment: number analyzed (Participants) | 11
  Dopamine concentration at 12 months off treatment | 6.43 [2.20 to 486.46]
  Dopamine concentration at 24 months off treatment: number analyzed (Participants) | 14
  Dopamine concentration at 24 months off treatment | 4.46 [0.04 to 1093.28]
  Dopamine concentration at 36 months off treatment: number analyzed (Participants) | 5
  Dopamine concentration at 36 months off treatment | 4.05 [0.11 to 9.32]
  3,4-dihydroxyphenylacetic acid concentration at baseline: number analyzed (Participants) | 15
  3,4-dihydroxyphenylacetic acid concentration at baseline | 2.56 [0.91 to 11.24]
  3,4-dihydroxyphenylacetic acid concentration at completion of treatment: number analyzed (Participants) | 14
  3,4-dihydroxyphenylacetic acid concentration at completion of treatment | 1.62 [0.82 to 9.91]
  3,4-dihydroxyphenylacetic acid concentration at 12 months off treatment: number analyzed (Participants) | 15
  3,4-dihydroxyphenylacetic acid concentration at 12 months off treatment | 1.04 [0.51 to 6.55]
  3,4-dihydroxyphenylacetic acid concentration at 24 months off treatment: number analyzed (Participants) | 14
  3,4-dihydroxyphenylacetic acid concentration at 24 months off treatment | 1.52 [0.31 to 6.70]
  3,4-dihydroxyphenylacetic acid concentration at 36 months off treatment: number analyzed (Participants) | 9
  3,4-dihydroxyphenylacetic acid concentration at 36 months off treatment | 1.00 [0.38 to 3.10]
  Hydroxytryptamine concentration at baseline: number analyzed (Participants) | 14
  Hydroxytryptamine concentration at baseline | 2.38 [0.12 to 13.94]
  Hydroxytryptamine concentration at completion of treatment: number analyzed (Participants) | 13
  Hydroxytryptamine concentration at completion of treatment | 2.01 [0.06 to 15.01]
  Hydroxytryptamine concentration at 12 months off treatment | 2.00 [0.06 to 8.46]
  Hydroxytryptamine concentration at 24 months off treatment: number analyzed (Participants) | 16
  Hydroxytryptamine concentration at 24 months off treatment | 2.44 [1.01 to 7.70]
  Hydroxytryptamine concentration at 36 months off treatment: number analyzed (Participants) | 9
  Hydroxytryptamine concentration at 36 months off treatment | 1.62 [0.29 to 8.85]
  Hydroxyindoleacetic acid concentration at baseline | 52.03 [30.02 to 400.35]
  Hydroxyindoleacetic acid concentration at completion of treatment | 52.72 [27.42 to 110.24]
  Hydroxyindoleacetic acid concentration at 12 months off treatment | 35.72 [24.58 to 51.60]
  Hydroxyindoleacetic acid concentration at 24 months off treatment | 33.98 [25.69 to 45.63]
  Hydroxyindoleacetic acid concentration at 36 months off treatment: number analyzed (Participants) | 9
  Hydroxyindoleacetic acid concentration at 36 months off treatment | 31.56 [16.09 to 53.04]
  Homovanillic acid concentration at baseline | 82.44 [34.57 to 565.30]
  Homovanillic acid concentration at completion of treatment | 114.13 [73.43 to 179.21]
  Homovanillic acid concentration at 12 months off treatment | 68.28 [40.78 to 146.84]
  Homovanillic acid concentration at 24 months off treatment | 88.27 [55.27 to 166.99]
  Homovanillic acid concentration at 36 months off treatment: number analyzed (Participants) | 9
  Homovanillic acid concentration at 36 months off treatment | 79.78 [35.40 to 152.51]

17. Secondary Outcome: Number and Type of Genetic Polymorphisms
Description: Types of genetic polymorphisms of neurotransmitters were examined. We studied 3 genetic polymorphisms; these were types of genetic polymorphisms involved in dopamine metabolism. They were as follows: rs6323, rs4680, and rs6280.
Time Frame: At study enrollment (Day 0)
Population: Three genetic polymorphisms involved in dopamine metabolism (rs6323, rs4680, and rs6280) were studied in 17 patients with CNS neurotransmitter studies.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Patients With Neurotransmitter Studies: Number of patients with neurotransmitter studies
Arm/Group | Number of Patients With Neurotransmitter Studies
Number analyzed (Participants) | 17
Participants
  rs6323 | 17
  rs4680 | 17
  rs6280 | 17

18. Secondary Outcome: Pharmacogenetic Variation on Central Nervous System Transmitters
Description: Frequencies of genetic polymorphisms were reported.
Time Frame: At study enrollment (Day 0)
Population: Eligible patients who had neurotransmitter studies performed. Seventeen patients had studies performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Neurotransmitter Studies
Number analyzed (Participants) | 17
Participants
  Genetic Polymorphisms for monoamine oxidase A (MAOA) rs6323: AA | 0
  Genetic Polymorphisms for monoamine oxidase A (MAOA) rs6323: AG | 0
  Genetic Polymorphisms for monoamine oxidase A (MAOA) rs6323: CC | 0
  Genetic Polymorphisms for monoamine oxidase A (MAOA) rs6323: GG | 2
  Genetic Polymorphisms for monoamine oxidase A (MAOA) rs6323: TC | 0
  Genetic Polymorphisms for monoamine oxidase A (MAOA) rs6323: TG | 2
  Genetic Polymorphisms for monoamine oxidase A (MAOA) rs6323: TT | 13
  Genetic Polymorphisms for catecholamine-O-methyltransferase (COMT) rs4680: AA | 5
  Genetic Polymorphisms for catecholamine-O-methyltransferase (COMT) rs4680: AG | 7
  Genetic Polymorphisms for catecholamine-O-methyltransferase (COMT) rs4680: CC | 0
  Genetic Polymorphisms for catecholamine-O-methyltransferase (COMT) rs4680: GG | 5
  Genetic Polymorphisms for catecholamine-O-methyltransferase (COMT) rs4680: TC | 0
  Genetic Polymorphisms for catecholamine-O-methyltransferase (COMT) rs4680: TG | 0
  Genetic Polymorphisms for catecholamine-O-methyltransferase (COMT) rs4680: TT | 0
  Genetic Polymorphisms for dopamine receptor D (DRD3) rs6280: AA | 0
  Genetic Polymorphisms for dopamine receptor D (DRD3) rs6280: AG | 0
  Genetic Polymorphisms for dopamine receptor D (DRD3) rs6280: CC | 6
  Genetic Polymorphisms for dopamine receptor D (DRD3) rs6280: GG | 0
  Genetic Polymorphisms for dopamine receptor D (DRD3) rs6280: TC | 4
  Genetic Polymorphisms for dopamine receptor D (DRD3) rs6280: TG | 0
  Genetic Polymorphisms for dopamine receptor D (DRD3) rs6280: TT | 7

19. Secondary Outcome: Number of Participants With Endocrinopathy
Description: Endocrine screening and growth hormone (GH) testing were done in consenting intermediate risk patients at the end of induction therapy, the end of all therapy, and at 6, 12, 24, 36, 48, and 60 months off therapy. Endocrinopathy was defined as the presence of central hypothyroidism (free T4 concentration below normal with low or normal TSH concentration), growth hormone deficiency (peak growth hormone concentration below 5 ng/mL on dynamic testing), or ACTH deficiency (cortisol concentration below 14 ug/dL after low dose cosyntropin stimulation). Numbers of participants with endocrinopathy at each time point are reported. Please note the small numbers of participants with available data.
Time Frame: End of induction therapy (approximately 16 weeks from start of treatment), end of therapy (approximately 48 weeks from start of treatment), and 6, 12, 24, 36, 48, and 60 months off therapy
Population: Endocrine screening and growth hormone (GH) testing were done in consenting intermediate risk patients.
Measure: Number; unit: participants
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 0 | 24 | 0
participants
  End of induction-number with endocrinopathy: number analyzed (Participants) | 0 | 13 | 0
  End of induction-number with endocrinopathy |  | 0 |
  End of therapy-number with endocrinopathy: number analyzed (Participants) | 0 | 8 | 0
  End of therapy-number with endocrinopathy |  | 0 |
  6-months off therapy-number with endocrinopathy: number analyzed (Participants) | 0 | 3 | 0
  6-months off therapy-number with endocrinopathy |  | 0 |
  12-months off therapy-number with endocrinopathy: number analyzed (Participants) | 0 | 1 | 0
  12-months off therapy-number with endocrinopathy |  | 0 |
  24-months off therapy-number with endocrinopathy: number analyzed (Participants) | 0 | 6 | 0
  24-months off therapy-number with endocrinopathy |  | 2 |
  36-months off therapy-number with endocrinopathy: number analyzed (Participants) | 0 | 1 | 0
  36-months off therapy-number with endocrinopathy |  | 0 |
  48-months off therapy-number with endocrinopathy: number analyzed (Participants) | 0 | 1 | 0
  48-months off therapy-number with endocrinopathy |  | 0 |
  60-months off therapy-number with endocrinopathy: number analyzed (Participants) | 0 | 1 | 0
  60-months off therapy-number with endocrinopathy |  | 1 |

20. Secondary Outcome: Growth Hormone Secretion
Description: Growth hormone secretion was measured in consenting intermediate risk patients at the end of induction therapy, the end of all therapy, and at 6, 12, 24, 36, 48, and 60 months off therapy. Mean growth hormone secretion values are reported by assessment time point. Please note the small numbers of participants with available data.
Time Frame: as for outcome 19
Population: Growth hormone secretion was measured in consenting intermediate risk patients. No Intermediate Risk patients had data available at 12, 36, 48, and 60 months off therapy.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 0 | 20 | 0
ng/mL
  End of induction: number analyzed (Participants) | 0 | 10 | 0
  End of induction |  | 15.3 (9.7) |
  End of therapy: number analyzed (Participants) | 0 | 8 | 0
  End of therapy |  | 13.4 (6.2) |
  6-months off therapy: number analyzed (Participants) | 0 | 2 | 0
  6-months off therapy |  | 7.3 (2.9) |
  12-months off therapy: number analyzed (Participants) | 0 | 0 | 0
  24-months off therapy: number analyzed (Participants) | 0 | 6 | 0
  24-months off therapy |  | 9.2 (6.5) |
  36-months off therapy: number analyzed (Participants) | 0 | 0 | 0
  48-months off therapy: number analyzed (Participants) | 0 | 0 | 0
  60-months off therapy: number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Methotrexate Clearance in Induction Cycle 1
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 1. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of Methotrexate (MTX)
Population: Eligible patients who received methotrexate during induction cycle 1 and had samples collected for PK analysis
Measure: Median (Full Range); unit: L/h/m^2
Groups:
- Low-Risk Group: Patients with gross total resection (GTR)/no evidence of metastatic disease (M0) medulloblastoma, nodular desmoplastic histology, or high grade glioma
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 37 | 94 | 44
L/h/m^2 | 5.69 [2.19 to 11.08] | 6.06 [3.07 to 10.69] | 5.65 [1.71 to 9.45]

22. Secondary Outcome: Methotrexate Clearance in Induction Cycle 2
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 2. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 93 | 41
L/h/m^2 | 5.47 [2.43 to 10.56] | 5.70 [2.71 to 8.98] | 5.70 [2.78 to 8.79]

23. Secondary Outcome: Methotrexate Clearance in Induction Cycle 3
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 3. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 3 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 35 | 82 | 36
L/h/m^2 | 5.68 [1.93 to 9.61] | 5.78 [2.59 to 9.27] | 5.81 [2.78 to 10.20]

24. Secondary Outcome: Methotrexate Clearance in Induction Cycle 4
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 4. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 4 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 34 | 80 | 34
L/h/m^2 | 5.75 [2.14 to 9.65] | 5.89 [2.95 to 8.84] | 5.79 [2.36 to 9.16]

25. Secondary Outcome: Methotrexate Volume of Central Compartment in Induction Cycle 1
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 1. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate volume of central compartment are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 37 | 94 | 44
L/m^2 | 11.63 [7.09 to 29.58] | 13.70 [7.03 to 28.21] | 13.25 [5.65 to 20.89]

26. Secondary Outcome: Methotrexate Volume of Central Compartment in Induction Cycle 2
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 2. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate volume of central compartment are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 93 | 41
L/m^2 | 13.77 [5.88 to 28.19] | 13.73 [6.47 to 31.45] | 13.62 [6.87 to 22.39]

27. Secondary Outcome: Methotrexate Volume of Central Compartment in Induction Cycle 3
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 3. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate volume of central compartment are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 3 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 35 | 82 | 36
L/m^2 | 12.70 [6.27 to 28.90] | 13.55 [7.31 to 24.48] | 13.87 [6.84 to 22.88]

28. Secondary Outcome: Methotrexate AUC0-66h in Induction Cycle 1
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 1. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate AUC0-66h (area under concentration curve from time 0 to 66 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 37 | 94 | 44
µmol·h/L | 1797 [993 to 5029] | 1813 [1029 to 3584] | 1821 [1053 to 3631]

29. Secondary Outcome: Methotrexate AUC0-66h in Induction Cycle 2
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 2. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate AUC0-66h (area under concentration curve from time 0 to 66 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 93 | 41
µmol·h/L | 1900 [1042 to 3267] | 1902 [1225 to 3742] | 1879 [1229 to 3271]

30. Secondary Outcome: Methotrexate Volume of Central Compartment in Induction Cycle 4
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 4. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate volume of central compartment are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 4 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 34 | 80 | 34
L/m^2 | 12.64 [7.16 to 22.92] | 13.31 [7.93 to 21.51] | 13.68 [6.94 to 21.82]

31. Secondary Outcome: Methotrexate AUC0-66h in Induction Cycle 3
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 3. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate AUC0-66h (area under concentration curve from time 0 to 66 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 3 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 35 | 82 | 36
µmol·h/L | 1872 [1145 to 3501] | 1879 [1187 to 3756] | 1831 [979 to 3139]

32. Secondary Outcome: Methotrexate AUC0-66h in Induction Cycle 4
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 4. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate AUC0-66h (area under concentration curve from time 0 to 66 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion and 6, 23, 42, 66 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 4 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 34 | 80 | 34
µmol·h/L | 1804 [1141 to 3504] | 1841 [1245 to 3727] | 1886 [1219 to 3491]

33. Secondary Outcome: Methotrexate Concentration at 42 Hours Post-dose in Induction Cycle 1
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 1. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate concentration at 42 hours post-dose are obtained using post hoc analysis.
Time Frame: 42 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 37 | 93 | 44
µmol/L | 0.49 [0.22 to 3.68] | 0.57 [0.15 to 4.61] | 0.61 [0.14 to 2.09]

34. Secondary Outcome: Methotrexate Concentration at 42 Hours Post-dose in Induction Cycle 2
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 2. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate concentration at 42 hours post-dose are obtained using post hoc analysis.
Time Frame: 42 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 93 | 41
µmol/L | 0.75 [0.19 to 3.09] | 0.72 [0.26 to 7.61] | 0.69 [0.24 to 1.49]

35. Secondary Outcome: Methotrexate Concentration at 42 Hours Post-dose in Induction Cycle 3
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 3. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate concentration at 42 hours post-dose are obtained using post hoc analysis.
Time Frame: 42 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 3 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 35 | 82 | 36
µmol/L | 0.65 [0.20 to 2.88] | 0.70 [0.16 to 4.34] | 0.58 [0.24 to 1.96]

36. Secondary Outcome: Methotrexate Concentration at 42 Hours Post-dose in Induction Cycle 4
Description: Methotrexate plasma concentration-time data are collected after the start of methotrexate infusion in induction cycle 4. Population parameters and inter-subject variability are estimated. Individual estimates of methotrexate concentration at 42 hours post-dose are obtained using post hoc analysis.
Time Frame: 42 hours from start of MTX
Population: Eligible patients who received methotrexate during induction cycle 4 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 34 | 80 | 34
µmol/L | 0.64 [0.26 to 3.12] | 0.64 [0.22 to 3.22] | 0.55 [0.20 to 1.79]

37. Secondary Outcome: Cyclophosphamide Clearance in Induction Chemotherapy
Description: Cyclophosphamide plasma concentration-time data are collected on day 9 in one cycle of induction chemotherapy. Individual estimates of cyclophosphamide clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during a cycle of induction therapy and had samples collected for PK analysis..
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 91 | 42
L/h/m^2 | 2.40 [1.16 to 9.15] | 2.23 [1.23 to 8.95] | 2.25 [0.84 to 3.40]

38. Secondary Outcome: Cyclophosphamide Clearance in Consolidation Chemotherapy Cycle 1
Description: Cyclophosphamide plasma concentration-time data are collected in consolidation cycle 1. Individual estimates of cyclophosphamide clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 20 | 4 | 28
L/h/m^2 | 2.39 [1.65 to 3.44] | 2.08 [1.97 to 2.62] | 2.43 [1.29 to 3.21]

39. Secondary Outcome: Cyclophosphamide Clearance in Consolidation Chemotherapy Cycle 2
Description: Cyclophosphamide plasma concentration-time data are collected in consolidation cycle 2. Individual estimates of cyclophosphamide clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 18 | 3 | 29
L/h/m^2 | 2.48 [1.97 to 3.35] | 2.55 [2.19 to 2.93] | 2.37 [1.61 to 3.16]

40. Secondary Outcome: Cyclophosphamide Apparent Oral Clearance in Maintenance Chemotherapy Cycle A1
Description: Cyclophosphamide plasma concentration-time data are collected on day 1 of maintenance cycle A1. Individual estimates of cyclophosphamide apparent oral clearance are obtained using post hoc analysis.
Time Frame: Pre-dose, 0.5, 1.75, 3 and 6 hours post-dose
Population: Eligible patients who received cyclophosphamide during maintenance cycle A1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 26 | 42 | 14
L/h/m^2 | 2.95 [2.05 to 3.89] | 2.83 [2.23 to 5.14] | 2.74 [2.23 to 4.02]

41. Secondary Outcome: Cyclophosphamide AUC0-24h in Induction Chemotherapy
Description: Cyclophosphamide plasma concentration-time data are collected on day 9 in one cycle of induction chemotherapy. Individual estimates of cyclophosphamide AUC0-24h (area under concentration curve from time 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: as for outcome 37
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 91 | 42
µmol·h/L | 2070 [592 to 4158] | 2150 [615 to 3430] | 2105 [1523 to 5121]

42. Secondary Outcome: Cyclophosphamide AUC0-24h in Consolidation Chemotherapy Cycle 1
Description: Cyclophosphamide plasma concentration-time data are collected in consolidation cycle 1. Individual estimates of cyclophosphamide AUC0-24h (area under concentration curve from time 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 20 | 4 | 28
µmol·h/L | 1968 [1480 to 2869] | 1504 [617 to 2511] | 868 [660 to 1498]

43. Secondary Outcome: 4-OH Cyclophosphamide AUC0-24h in Consolidation Chemotherapy Cycle 1
Description: 4-OH cyclophosphamide plasma concentration-time data are collected in consolidation cycle 1. Individual estimates of 4-OH cyclophosphamide AUC0-24h (area under concentration curve from time 0 to 24 hours post- dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 20 | 4 | 28
µmol·h/L | 96.8 [63.0 to 124.4] | 48.7 [25.8 to 124.6] | 39.8 [25.5 to 59.8]

44. Secondary Outcome: Cyclophosphamide AUC0-24h in Consolidation Chemotherapy Cycle 2
Description: Cyclophosphamide plasma concentration-time data are collected in consolidation cycle 2. Individual estimates of cyclophosphamide AUC0-24h (area under concentration curve from time 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 18 | 3 | 29
µmol·h/L | 1966 [1437 to 2519] | 799 [740 to 2303] | 899 [700 to 1240]

45. Secondary Outcome: Cyclophosphamide AUC0-24h in Maintenance Chemotherapy Cycle A1
Description: Cyclophosphamide plasma concentration-time data are collected on day 1 of maintenance cycle A1. Individual estimates of cyclophosphamide AUC0-24h are obtained using post hoc analysis.
Time Frame: Pre-dose, 0.5, 1.75, 3, 6, and 24 hours post-dose
Population: Eligible patients who received cyclophosphamide during maintenance cycle A1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 26 | 42 | 14
µmol·h/L | 39.9 [25.3 to 51.3] | 38.7 [21.2 to 54.9] | 42.2 [28.0 to 53.0]

46. Secondary Outcome: 4-OH Cyclophosphamide AUC0-24h in Induction Chemotherapy
Description: 4-OH cyclophosphamide plasma concentration-time data are collected on day 9 in one cycle of induction chemotherapy. Individual estimates of 4-OH cyclophosphamide AUC0-24h (area under concentration curve from time 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: as for outcome 37
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 91 | 42
µmol·h/L | 116.4 [74.6 to 200.3] | 111.3 [71.4 to 181.0] | 109.1 [65.0 to 175.0]

47. Secondary Outcome: 4-OH Cyclophosphamide AUC0-24h in Consolidation Chemotherapy Cycle 2
Description: 4-OH cyclophosphamide plasma concentration-time data are collected in consolidation cycle 2. Individual estimates of 4-OH cyclophosphamide AUC0-24h (area under concentration curve from time 0 to 24 hours post- dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 18 | 3 | 29
µmol·h/L | 95.9 [81.7 to 131.1] | 49.5 [39.5 to 84.5] | 43.5 [30.8 to 72.5]

48. Secondary Outcome: 4-OH Cyclophosphamide AUC0-24h in Maintenance Chemotherapy Cycle A1
Description: 4-OH cyclophosphamide plasma concentration-time data are collected on day 1 of maintenance cycle A1. Individual estimates of 4-OH cyclophosphamide AUC0-24h (area under concentration curve from time 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-dose, 0.5, 1.75, 3, 6, and 24 hours post-dose
Population: Eligible patients who received cyclophosphamide during maintenance cycle A1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 26 | 42 | 14
µmol·h/L | 1.98 [0.98 to 3.01] | 1.96 [1.12 to 3.08] | 1.82 [1.19 to 2.40]

49. Secondary Outcome: CEPM AUC0-24h in Induction Chemotherapy
Description: Carboxyethylphosphoramide mustard (CEPM) plasma concentration-time data are collected on day 9 in one induction cycle. Individual estimates of CEPM AUC0-24h (area under concentration curve from time 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: as for outcome 37
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 38 | 91 | 42
µmol·h/L | 140.2 [50.1 to 453.0] | 137.8 [80.4 to 328.9] | 135.3 [57.6 to 591.7]

50. Secondary Outcome: CEPM AUC0-24h in Consolidation Chemotherapy Cycle 1
Description: Carboxyethylphosphoramide mustard (CEPM) plasma concentration-time data are collected in consolidation cycle 1. Individual estimates of CEPM AUC0-24h (area under concentration curve from time 0 to 24 hours post- dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 20 | 4 | 28
µmol·h/L | 128.9 [90.8 to 272.9] | 62.2 [48.8 to 193.9] | 51.8 [18.9 to 97.0]

51. Secondary Outcome: CEPM AUC0-24h in Consolidation Chemotherapy Cycle 2
Description: Carboxyethylphosphoramide mustard (CEPM) plasma concentration-time data are collected in consolidation cycle 2. Individual estimates of CEPM AUC0-24h (area under concentration curve from time 0 to 24 hours post- dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, end of infusion, 3, 6, and 24 hours from end of cyclophosphamide infusion
Population: Eligible patients who received cyclophosphamide during consolidation cycle 2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 18 | 3 | 29
µmol·h/L | 132.7 [89.7 to 244.0] | 46.8 [41.9 to 69.0] | 44.0 [21.1 to 73.9]

52. Secondary Outcome: CEPM AUC0-24h in Maintenance Chemotherapy Cycle A1
Description: Carboxyethylphosphoramide mustard (CEPM) plasma concentration-time data are collected on day 1 of maintenance cycle A1. Individual estimates of CEPM AUC0-24h (area under concentration curve from time 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-dose, 0.5, 1.75, 3, 6, and 24 hours post-dose
Population: Eligible patients who received cyclophosphamide during maintenance cycle A1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 26 | 42 | 14
µmol·h/L | 1.59 [0.75 to 3.48] | 1.65 [0.68 to 3.64] | 1.41 [0.64 to 3.96]

53. Secondary Outcome: Participants With Empirical Dosage Achieving Target System Exposure of Intravenous Topotecan
Description: Number of participants who successfully achieve target systemic exposure of intravenous topotecan after an empiric dosage during consolidation phase of therapy are reported.
Time Frame: Pre-infusion, 5 min., 1, and 3 hours from end of infusion
Population: Eligible patients who received topotecan with empirical dosage during consolidation therapy were included in this analysis. Per protocol, low-risk and intermediate-risk patients did not receive topotecan during consolidation unless they experienced disease progression during induction. One such intermediate-risk patient was included.
Measure: Number; unit: participants
Arm/Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 1 | 27
participants | 0 | 8

54. Secondary Outcome: Participants With PK-guided Dosage Adjustment Achieving Target System Exposure of Intravenous Topotecan
Description: Number of participants who successfully achieve target systemic exposure of intravenous topotecan after a pharmacokinetic-guided dosage adjustment during consolidation phase of therapy are reported.
Time Frame: Pre-infusion, 5 min., 1, and 3 hours from end of infusion
Population: Eligible patients who received topotecan with PK-guided dosage adjustment during consolidation therapy were included in this analysis. Per protocol, low-risk and intermediate-risk patients did not receive topotecan during consolidation unless they experienced disease progression during induction. One such intermediate-risk patient was included.
Measure: Number; unit: participants
Arm/Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 1 | 27
participants | 1 | 20

55. Secondary Outcome: Topotecan Clearance in Consolidation Chemotherapy
Description: Topotecan plasma concentration-time data are collected on day 1 of consolidation cycle 1 after a single IV dose. Individual estimates of topotecan clearance are obtained using post hoc analysis.
Time Frame: Pre-infusion, 5 min., 1, and 3 hours from end of infusion
Population: Eligible patients who received intravenous topotecan during consolidation cycle 1 and had PK samples collected were included in this analysis. Per protocol, low- and intermediate-risk patients did not receive topotecan during consolidation unless they experienced disease progression during induction. One such intermediate-risk patient was included.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 1 | 27
L/h/m^2 | 30.3 [30.3 to 30.3] | 26.40 [6.8 to 43.0]

56. Secondary Outcome: Topotecan Apparent Oral Clearance in Maintenance Chemotherapy
Description: Topotecan plasma concentration-time data are collected on day 1 of maintenance cycle A1 after a single oral dose. Individual estimates of topotecan apparent oral clearance are obtained using post hoc analysis.
Time Frame: Pre-dose, 0.25, 1.5 and 6 hours post-dose
Population: Eligible patients who received oral topotecan during maintenance therapy cycle A1 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 18 | 33 | 10
L/h | 41.4 [12.3 to 54.6] | 41.0 [24.4 to 62.7] | 44.6 [18.1 to 57.0]

57. Secondary Outcome: Topotecan AUC0-24h in Consolidation Chemotherapy
Description: Topotecan plasma concentration-time data are collected on day 1 of consolidation cycle 1 after a single IV dose. Individual estimates of topotecan AUC0-24h (area under concentration curve from time 0 to 24 hours post- dose) are obtained using post hoc analysis.
Time Frame: Pre-infusion, 5 min., 1, 3, and 24 hours from end of infusion
Population: as for outcome 55
Measure: Median (Full Range); unit: µg·h/L
Arm/Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 1 | 27
µg·h/L | 117 [117 to 117] | 116 [90 to 262]

58. Secondary Outcome: Topotecan AUC0-24h in Maintenance Chemotherapy
Description: Topotecan plasma concentration-time data are collected on day 1 of maintenance cycle A1 after a single oral dose. Individual estimates of topotecan AUC0-24h (area under concentration curve from time 0 to 24 hours post- dose) are obtained using post hoc analysis.
Time Frame: Pre-dose, 0.25, 1.5, 6, and 24 hours post-dose
Population: as for outcome 56
Measure: Median (Full Range); unit: µg·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 18 | 33 | 10
µg·h/L | 10.90 [9.04 to 24.36] | 11.60 [7.93 to 20.50] | 10.33 [7.96 to 16.61]

59. Secondary Outcome: Erlotinib Apparent Oral Clearance
Description: Erlotinib plasma concentration-time data are collected on day 1 of maintenance cycle B2. Individual estimates of erlotinib apparent oral clearance are obtained using post hoc analysis.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose
Population: Eligible patients who received oral erlotinib during maintenance therapy cycle B2 and had samples collected for PK analysis.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 10 | 11 | 3
L/h/m^2 | 6.53 [3.13 to 18.55] | 7.79 [3.87 to 16.84] | 8.40 [5.96 to 10.46]

60. Secondary Outcome: Erlotinib Apparent Volume of Central Compartment
Description: Erlotinib plasma concentration-time data are collected on day 1 of maintenance cycle B2. Individual estimates of erlotinib apparent volume of central compartment are obtained using post hoc analysis.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose
Population: as for outcome 59
Measure: Median (Full Range); unit: L/m^2
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 10 | 11 | 3
L/m^2 | 72.9 [39.5 to 233.7] | 61.7 [41.3 to 119.0] | 104.8 [47.6 to 109.9]

61. Secondary Outcome: Erlotinib AUC0-24h
Description: Erlotinib plasma concentration-time data are collected on day 1 of maintenance cycle B2. Individual estimates of erlotinib AUC0-24h (area under concentration curve from 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose
Population: as for outcome 59
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 10 | 11 | 3
µmol·h/L | 31.0 [7.2 to 64.8] | 23.5 [12.5 to 48.6] | 22.0 [13.8 to 33.0]

62. Secondary Outcome: OSI-420 AUC0-24h
Description: Erlotinib metabolite OSI-420 plasma concentration-time data are collected on day 1 of maintenance cycle B2. Individual estimates of OSI-420 AUC0-24h (area under concentration curve from 0 to 24 hours post-dose) are obtained using post hoc analysis.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose
Population: as for outcome 59
Measure: Median (Full Range); unit: µmol·h/L
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 10 | 11 | 3
µmol·h/L | 2.17 [0.73 to 5.98] | 1.81 [1.17 to 6.97] | 1.62 [1.25 to 2.93]

63. Secondary Outcome: Rate of Local Disease Progression
Description: Local failure was defined as the interval from end of RT to date of local failure (or combined local + distant failure). Competing events were distant failure or second malignancy. Patients without an event were censored at date of last contact. The 1-year cumulative incidence was estimated and reported with a 95% confidence interval.
Time Frame: 1 year after completion of radiation therapy for last patient
Population: Eligible intermediate-risk patients who received focal radiation were included in this analysis. Of the 156 intermediate risk patients, 121 started radiation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Intermediate-risk Patients Who Received Focal Radiation: Patients with no evidence of metastatic disease (M0) medulloblastoma or nodular desmoplastic histology with less than a surgical gross total resection (GTR), other histologic diagnoses with no metastatic disease who received induction chemotherapy and intermediate-risk therapy that included focal radiation.
Arm/Group | Intermediate-risk Patients Who Received Focal Radiation
Number analyzed (Participants) | 121
Percentage of participants | 13.2 [7.2 to 19.3]

64. Secondary Outcome: Rate of Distant Disease Progression
Description: Distant failure was defined as the interval from end of RT to date of distant failure (or combined local + distant failure). Competing events were local failure or second malignancy. Patients without an event were censored at date of last contact. The 1-year cumulative incidence was estimated and reported with a 95% confidence interval.
Time Frame: 1 year after completion of radiation therapy for last patient
Population: as for outcome 63
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Intermediate-risk Patients Who Received Focal Radiation: Patients with M0 medulloblastoma or nodular desmoplastic histology with less than a GTR, other histologic diagnoses with no metastatic disease who received induction chemotherapy and intermediate-risk therapy that included focal radiation.
Arm/Group | Intermediate-risk Patients Who Received Focal Radiation
Number analyzed (Participants) | 121
percentage of participants | 25.6 [17.8 to 33.4]

65. Secondary Outcome: Neurocognitive Performance Related to Global Cognitive Functioning as Measured by Cognitive Composite Scores and Estimated IQ Scores
Description: Global cognitive functioning was measured based on Cognitive Composite Scores from the Bayley III instrument for subjects <3 years of age and on estimated IQ scores from the Stanford Binet V instrument for subjects ≥3 years of age. Higher scores indicate better performance. The normative mean is 100 with a standard deviation of 15.
Time Frame: Baseline, prior to maintenance therapy, completion of therapy, and 12 months, 24 months, 36 months, 48 months, and 60 months off therapy
Population: Eligible patients with scores at any of the data collection timepoints were included. Sample sizes differ across timepoints as not all subjects had scores for all timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 48 | 111 | 41
score on a scale
  Baseline: number analyzed (Participants) | 39 | 87 | 38
  Baseline | 88.6 (17.6) | 91.0 (15.4) | 87.4 (22.3)
  Prior to Maintenance Therapy: number analyzed (Participants) | 33 | 64 | 18
  Prior to Maintenance Therapy | 91.1 (16.8) | 92.3 (15.1) | 94.8 (19.0)
  Completion of Therapy: number analyzed (Participants) | 28 | 44 | 9
  Completion of Therapy | 85.8 (17.5) | 93.4 (15.3) | 76.8 (18.6)
  12 Months Off Therapy: number analyzed (Participants) | 23 | 35 | 9
  12 Months Off Therapy | 89.2 (21.3) | 89.9 (15.6) | 83.3 (18.3)
  24 Months Off Therapy: number analyzed (Participants) | 15 | 36 | 6
  24 Months Off Therapy | 97.6 (16.7) | 89.4 (19.0) | 77.7 (21.0)
  36 Months Off Therapy: number analyzed (Participants) | 14 | 31 | 4
  36 Months Off Therapy | 92.4 (26.0) | 89.9 (16.2) | 81.3 (17.4)
  48 Months Off Therapy: number analyzed (Participants) | 15 | 30 | 6
  48 Months Off Therapy | 85.3 (24.1) | 91.3 (18.4) | 85.2 (27.4)
  60 Months Off Therapy: number analyzed (Participants) | 15 | 22 | 4
  60 Months Off Therapy | 82.0 (25.6) | 85.3 (17.9) | 71.5 (18.4)

66. Secondary Outcome: Neurocognitive Performance Related to Attention as Measured by Attention Problems T-scores
Description: Scores measuring attention were obtained from the Attention Problems T-score on the BASC-2 instrument which is a parent report. Higher scores indicate more attention problems. The normative mean is 50 with a standard deviation of 10.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 40 | 86 | 34
score on a scale
  Baseline: number analyzed (Participants) | 13 | 47 | 22
  Baseline | 51.7 (10.9) | 49.6 (9.5) | 49.2 (9.1)
  Prior to Maintenance Therapy: number analyzed (Participants) | 12 | 43 | 9
  Prior to Maintenance Therapy | 53.5 (9.5) | 51.3 (9.9) | 52.4 (4.6)
  Completion of Therapy: number analyzed (Participants) | 17 | 43 | 3
  Completion of Therapy | 52.6 (8.6) | 50.9 (9.4) | 43.3 (12.7)
  12 Months Off Therapy: number analyzed (Participants) | 22 | 41 | 9
  12 Months Off Therapy | 56.2 (10.1) | 53.9 (10.2) | 53.9 (13.0)
  24 Months Off Therapy: number analyzed (Participants) | 20 | 36 | 10
  24 Months Off Therapy | 54.5 (10.6) | 55.3 (10.1) | 49.8 (12.6)
  36 Months Off Therapy: number analyzed (Participants) | 15 | 33 | 6
  36 Months Off Therapy | 53.3 (8.3) | 55.1 (9.8) | 53.3 (12.2)
  48 Months Off Therapy: number analyzed (Participants) | 16 | 31 | 6
  48 Months Off Therapy | 56.4 (10.4) | 55.5 (10.1) | 55.3 (10.3)
  60 Months Off Therapy: number analyzed (Participants) | 16 | 22 | 5
  60 Months Off Therapy | 51.9 (11.5) | 57.7 (12.0) | 58.8 (12.5)

67. Secondary Outcome: Neurocognitive Performance Related to Processing Speed as Measured by Visual Matching Standard Scores
Description: Scores measuring processing speed were obtained based on the visual matching standard score from the Woodcock Johnson III instrument. Higher scores indicate better performance. The normative mean is 100 with a standard deviation of 15.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 23 | 49 | 9
score on a scale
  Baseline: number analyzed (Participants) | 1 | 6 | 1
  Baseline | 119.0 | 96.5 (11.0) | 107.0
  Prior to Maintenance Therapy: number analyzed (Participants) | 1 | 8 | 2
  Prior to Maintenance Therapy | 89.0 | 97.6 (12.3) | 109.5 (2.1)
  Completion of Therapy: number analyzed (Participants) | 4 | 13 | 0
  Completion of Therapy | 105.3 (20.2) | 100.2 (15.2) |
  12 Months Off Therapy: number analyzed (Participants) | 5 | 17 | 1
  12 Months Off Therapy | 96.8 (9.8) | 93.1 (13.3) | 71.0
  24 Months Off Therapy: number analyzed (Participants) | 12 | 26 | 3
  24 Months Off Therapy | 98.4 (16.6) | 90.2 (15.3) | 89.3 (13.3)
  36 Months Off Therapy: number analyzed (Participants) | 11 | 25 | 4
  36 Months Off Therapy | 101.6 (15.8) | 89.7 (20.2) | 89.8 (12.4)
  48 Months Off Therapy: number analyzed (Participants) | 13 | 26 | 3
  48 Months Off Therapy | 93.2 (23.9) | 87.6 (14.7) | 78.7 (17.0)
  60 Months Off Therapy: number analyzed (Participants) | 13 | 17 | 1
  60 Months Off Therapy | 86.3 (36.2) | 84.6 (17.1) | 65.0

68. Secondary Outcome: Neurocognitive Performance Related to Executive Functioning as Measured by Global Executive Composite T-scores
Description: Scores measuring executive functioning were obtained from Global Executive Composite (GEC) T-scores, which were obtained from the Behavior Rating Inventory of Executive Function (BRIEF) instrument which is a parent report. Higher scores indicate more problems. The normative mean is 50 with a standard deviation of 10.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 40 | 85 | 34
score on a scale
  Baseline: number analyzed (Participants) | 13 | 48 | 22
  Baseline | 59.2 (16.0) | 49.6 (9.7) | 52.4 (13.1)
  Prior to Maintenance Therapy: number analyzed (Participants) | 12 | 44 | 9
  Prior to Maintenance Therapy | 54.3 (9.9) | 52.5 (12.3) | 49.3 (11.9)
  Completion of Therapy: number analyzed (Participants) | 17 | 40 | 3
  Completion of Therapy | 55.3 (11.9) | 50.6 (10.1) | 45.3 (14.7)
  12 Months Off Therapy: number analyzed (Participants) | 22 | 39 | 9
  12 Months Off Therapy | 57.9 (13.7) | 56.5 (14.3) | 60.1 (20.0)
  24 Months Off Therapy: number analyzed (Participants) | 20 | 37 | 10
  24 Months Off Therapy | 59.9 (16.5) | 55.1 (13.6) | 52.1 (9.6)
  36 Months Off Therapy: number analyzed (Participants) | 15 | 32 | 6
  36 Months Off Therapy | 55.7 (12.8) | 57.7 (11.8) | 58.2 (11.1)
  48 Months Off Therapy: number analyzed (Participants) | 16 | 33 | 6
  48 Months Off Therapy | 60.3 (16.8) | 55.6 (11.7) | 49.5 (10.6)
  60 Months Off Therapy: number analyzed (Participants) | 15 | 21 | 5
  60 Months Off Therapy | 55.1 (11.8) | 58.3 (15.0) | 55.2 (13.4)

69. Secondary Outcome: Neurocognitive Performance Related to Working Memory as Measured by Working Memory T-scores
Description: Scores measuring working memory were obtained from Working Memory T-scores, which were obtained from the Behavior Rating Inventory of Executive Function (BRIEF) instrument which is a parent report. Higher scores indicate more problems. The normative mean is 50 with a standard deviation of 10.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 40 | 85 | 34
score on a scale
  Baseline: number analyzed (Participants) | 13 | 48 | 22
  Baseline | 63.2 (16.0) | 51.6 (10.8) | 57.0 (13.6)
  Prior to Maintenance Therapy: number analyzed (Participants) | 12 | 44 | 9
  Prior to Maintenance Therapy | 58.7 (10.7) | 55.5 (13.3) | 54.1 (11.1)
  Completion of Therapy: number analyzed (Participants) | 17 | 41 | 3
  Completion of Therapy | 60.8 (14.9) | 54.9 (11.1) | 49.0 (16.8)
  12 Months Off Therapy: number analyzed (Participants) | 22 | 39 | 9
  12 Months Off Therapy | 64.4 (16.1) | 60.4 (14.5) | 67.7 (22.3)
  24 Months Off Therapy: number analyzed (Participants) | 20 | 38 | 10
  24 Months Off Therapy | 63.6 (17.8) | 59.4 (14.7) | 55.4 (13.3)
  36 Months Off Therapy: number analyzed (Participants) | 15 | 32 | 6
  36 Months Off Therapy | 59.3 (13.9) | 62.0 (14.2) | 61.7 (8.6)
  48 Months Off Therapy: number analyzed (Participants) | 16 | 34 | 6
  48 Months Off Therapy | 60.9 (16.1) | 60.0 (13.1) | 54.5 (12.8)
  60 Months Off Therapy: number analyzed (Participants) | 16 | 21 | 5
  60 Months Off Therapy | 56.8 (13.3) | 60.6 (14.3) | 61.0 (15.3)

70. Secondary Outcome: Neurocognitive Performance Related to Verbal Fluency as Measured by Retrieval Fluency Standard Scores
Description: Scores measuring verbal fluency were obtained from Retrieval Fluency standard scores on the Woodcock Johnson III instrument. Higher scores indicate better performance. The normative mean is 100 with a standard deviation of 15.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 25 | 50 | 10
score on a scale
  Baseline: number analyzed (Participants) | 1 | 6 | 0
  Baseline | 117.0 | 87.7 (18.4) |
  Prior to Maintenance Therapy: number analyzed (Participants) | 2 | 9 | 0
  Prior to Maintenance Therapy | 97.0 (5.7) | 89.4 (13.4) |
  Completion of Therapy: number analyzed (Participants) | 4 | 14 | 0
  Completion of Therapy | 90.0 (13.2) | 95.3 (14.4) |
  12 Months Off Therapy: number analyzed (Participants) | 6 | 21 | 2
  12 Months Off Therapy | 94.8 (11.4) | 86.1 (19.9) | 87.0 (1.4)
  24 Months Off Therapy: number analyzed (Participants) | 10 | 26 | 4
  24 Months Off Therapy | 98.8 (9.7) | 82.5 (20.6) | 90.8 (4.6)
  36 Months Off Therapy: number analyzed (Participants) | 12 | 27 | 5
  36 Months Off Therapy | 100.2 (13.3) | 88.1 (24.9) | 81.4 (14.9)
  48 Months Off Therapy: number analyzed (Participants) | 13 | 25 | 3
  48 Months Off Therapy | 77.1 (16.0) | 88.7 (16.0) | 95.7 (15.0)
  60 Months Off Therapy: number analyzed (Participants) | 14 | 18 | 3
  60 Months Off Therapy | 81.9 (22.1) | 87.9 (16.4) | 70.3 (23.7)

71. Secondary Outcome: Neurocognitive Performance Related to Visual-spatial Reasoning as Measured by Visual Motor Integration (VMI) T-scores
Description: Scores measuring visual-spatial reasoning were obtained from VMI T-scores on the Beery VMI instrument. Higher scores indicate better performance. The normative mean is 50 with standard deviation of 10.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 27 | 53 | 14
score on a scale
  Baseline: number analyzed (Participants) | 1 | 11 | 3
  Baseline | 62.0 | 47.5 (16.3) | 37.3 (11.9)
  Prior to Maintenance Therapy: number analyzed (Participants) | 2 | 20 | 2
  Prior to Maintenance Therapy | 39.0 (17.0) | 44.6 (12.6) | 53.0 (0.0)
  Completion Of Therapy: number analyzed (Participants) | 4 | 17 | 1
  Completion Of Therapy | 40.0 (13.6) | 48.5 (8.6) | 46.0
  12 Months Off Therapy: number analyzed (Participants) | 11 | 26 | 3
  12 Months Off Therapy | 43.1 (18.2) | 43.8 (11.1) | 39.0 (9.2)
  24 Months Off Therapy: number analyzed (Participants) | 13 | 34 | 5
  24 Months Off Therapy | 48.2 (11.5) | 43.6 (10.3) | 32.0 (16.0)
  36 Months Off Therapy: number analyzed (Participants) | 13 | 29 | 5
  36 Months Off Therapy | 45.6 (14.1) | 41.3 (8.9) | 36.8 (13.6)
  48 Months Off Therapy: number analyzed (Participants) | 14 | 26 | 3
  48 Months Off Therapy | 44.2 (23.5) | 43.6 (7.3) | 44.3 (10.1)
  60 Months Off Therapy: number analyzed (Participants) | 16 | 19 | 3
  60 Months Off Therapy | 39.4 (16.7) | 40.6 (9.2) | 34.0 (15.7)

72. Secondary Outcome: Neurocognitive Performance Related to Visual-spatial Reasoning as Measured by Visual Perception T-scores
Description: Scores measuring visual-spatial reasoning were obtained from Visual Perception T-scores on the Beery Visual Motor Integration (VMI) instrument. Higher scores indicate better performance. The normative mean is 50 with a standard deviation of 10.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 22 | 53 | 14
score on a scale
  Baseline: number analyzed (Participants) | 1 | 9 | 3
  Baseline | 66.0 | 31.6 (12.2) | 33.7 (9.5)
  Prior to Maintenance Therapy: number analyzed (Participants) | 2 | 14 | 2
  Prior to Maintenance Therapy | 32.0 (7.1) | 40.2 (12.2) | 56.0 (8.5)
  Completion of Therapy: number analyzed (Participants) | 3 | 16 | 2
  Completion of Therapy | 39.0 (16.4) | 39.8 (12.3) | 18.5 (26.2)
  12 Months Off Therapy: number analyzed (Participants) | 6 | 21 | 1
  12 Months Off Therapy | 42.3 (14.7) | 41.0 (14.5) | 33.0
  24 Months Off Therapy: number analyzed (Participants) | 11 | 31 | 3
  24 Months Off Therapy | 43.4 (15.0) | 40.1 (13.4) | 32.0 (8.9)
  36 Months Off Therapy: number analyzed (Participants) | 11 | 26 | 5
  36 Months Off Therapy | 51.2 (17.8) | 41.0 (13.6) | 48.8 (18.7)
  48 Months Off Therapy: number analyzed (Participants) | 13 | 24 | 3
  48 Months Off Therapy | 48.6 (24.9) | 46.1 (11.3) | 42.7 (8.3)
  60 Months Off Therapy: number analyzed (Participants) | 14 | 19 | 2
  60 Months Off Therapy | 43.1 (18.8) | 42.3 (13.3) | 36.0 (12.7)

73. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in right frontal-lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-risk Group | Intermediate-risk Group | High-risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0019 [0.0016 to 0.0022] | 0.0016 [0.0015 to 0.0018] | 0.0017 [0.0015 to 0.0019]

74. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in left frontal lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
change in FA per month | 0.0019 [0.0015 to 0.0022] | 0.0017 [0.0015 to 0.0018] | 0.0017 [0.0014 to 0.0019]

75. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in right parietal lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0015 [0.0012 to 0.0019] | 0.0014 [0.0012 to 0.0015] | 0.0016 [0.0013 to 0.0018]

76. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in left parietal lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0016 [0.0012 to 0.002] | 0.0014 [0.0012 to 0.0016] | 0.0016 [0.0013 to 0.0018]

77. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in right occipital lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0016 [0.0013 to 0.0019] | 0.0015 [0.0014 to 0.0017] | 0.0013 [0.0011 to 0.0016]

78. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in left occipital lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0021 [0.0017 to 0.0025] | 0.0020 [0.0018 to 0.0022] | 0.0015 [0.0012 to 0.0018]

79. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in right temporal lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0014 [0.0012 to 0.0017] | 0.0013 [0.0011 to 0.0014] | 0.0013 [0.0011 to 0.0015]

80. Secondary Outcome: Change in Neurostructure, Especially White Matter Volume and Integrity
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in left temporal lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0014 [0.0011 to 0.0017] | 0.0013 [0.0011 to 0.0014] | 0.0014 [0.0011 to 0.0016]

81. Secondary Outcome: Change in Quantitative Magnetic Resonance (MR) Measures in the Frontal Lobe
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in frontal lobe over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0019 [0.0016 to 0.0022] | 0.0017 [0.0015 to 0.0018] | 0.0017 [0.0014 to 0.0019]

82. Secondary Outcome: Change in Quantitative MR Measures in the Right Frontal-parietal Regions
Description: Quantitative MRI measures Fractional Anisotropy (FA) change per month in right frontal-parietal region over time in each risk group will be assessed using a random effects model incorporating various covariates. Covariates to be considered include age at diagnosis, time since diagnosis and risk-arm. Differences in quantitative MRI measures of neurostructure volume and integrity between patient groups will be evaluated as a metric of structural neurotoxicity of therapy.
  Fractional anisotropy (FA) is a scalar unitless measure that quantifies the degree of anisotropy of a diffusion process, particularly in the context of diffusion tensor imaging (DTI) used in MRI scans. FA values range from 0 to 1
Time Frame: From baseline (month 0) to 60 months (therapy duration lasted approximately 48 weeks or 11 months)
Population: Eligible infratentorial medulloblastoma, ependymoma, and pineoblastoma patients(n=75) were included.
Measure: Number (95% Confidence Interval); unit: Change in FA per month
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
Number analyzed (Participants) | 12 | 43 | 20
Change in FA per month | 0.0017 [0.0014 to 0.0021] | 0.0015 [0.0014 to 0.0017] | 0.0016 [0.0014 to 0.0019]

ADVERSE EVENTS:
Time Frame: All adverse events grades 3, 4, and 5 which occur during treatment and for 30 days after the end of treatment, and events which occur later than 30 days after the end of treatment which are felt to be at least possibly related to treatment, to the time of off study, were collected with some exceptions noted in the additional description section, up to 6 years..
Description: Per protocol, some grade 3 and 4 hematologic toxicities, grade 3 elevation in serum ALT or AST, grade 3 and 4 electrolyte abnormalities, and total parenteral nutrition or intravenous fluids administered to prevent significant weight loss/malnutrition were not collected, especially if they occurred from the beginning of induction chemotherapy. The one patient in the high-risk group who did not start therapy due to early disease progression was excluded from adverse event results.
Arm/Group | Low-Risk Group | Intermediate-Risk Group | High-Risk Group
All-Cause Mortality (participants affected / at risk) | 10/57 | 58/156 | 49/77
Serious Adverse Events (participants affected / at risk) | 3/57 | 7/156 | 5/76
Other Adverse Events (participants affected / at risk) | 55/57 | 145/156 | 70/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Risk Group (N=57) | Intermediate-Risk Group (N=156) | High-Risk Group (N=76)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 3 (3) | 0 (0)
Weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Perforation, GI, Duodenum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), Pharynx (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Documented clinically or microbiologically
Infection, Upper airway NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, Blood (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, Catheter-related (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, Eye NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Irritability (children <3 years of age) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurology - Other (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils, Wound (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Risk Group (N=57) | Intermediate-Risk Group (N=156) | High-Risk Group (N=76)
Febrile neutropenia (Blood and lymphatic system disorders) | 36 (83) | 92 (169) | 48 (120) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 32 (60) | 57 (124) | 10 (20)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 24 (38) | 45 (83) | 6 (11)
Vomiting (Gastrointestinal disorders) | 10 (11) | 25 (32) | 22 (29)
Hemoglobin (Blood and lymphatic system disorders) | 13 (15) | 9 (20) | 3 (3)
Infection, Catheter-related (Infections and infestations) | 11 (14) | 17 (19) | 8 (9) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Anorexia (Gastrointestinal disorders) | 6 (7) | 15 (16) | 12 (13)
Infection with normal ANC or Grade 1 or 2 neutrophils, Catheter-related (Infections and infestations) | 8 (8) | 19 (26) | 5 (7)
Platelets (Blood and lymphatic system disorders) | 7 (19) | 8 (9) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (10) | 9 (13)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (7) | 8 (8) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 13 (14) | 8 (11)
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 4 (4) | 7 (8) | 7 (7)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 3 (3) | 8 (12) | 7 (10)
Infection, Skin (cellulitis) (Infections and infestations) | 0 (0) | 7 (9) | 7 (7) — Documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Seizure (Nervous system disorders) | 1 (1) | 4 (5) | 7 (7)
Infection, Blood (Infections and infestations) | 5 (5) | 5 (6) | 5 (5) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Weight loss (General disorders) | 1 (1) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 6 (6)
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 1 (1) | 11 (12) | 4 (5)
Infection - Other (Infections and infestations) | 4 (4) | 8 (11) | 4 (5)
Hydrocephalus (Nervous system disorders) | 2 (2) | 8 (9) | 5 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils, Blood (Infections and infestations) | 2 (3) | 9 (9) | 4 (4)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (4) | 8 (9) | 3 (3)
Infection, Upper airway NOS (Infections and infestations) | 1 (1) | 4 (4) | 4 (4) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Urinary tract NOS (Infections and infestations) | 1 (1) | 2 (3) | 4 (4) — Documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Lymphopenia (Blood and lymphatic system disorders) | 2 (6) | 8 (8) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 8 (8) | 3 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 8 (9) | 3 (3)

LIMITATIONS AND CAVEATS:
Results for the some of the secondary objectives are not available yet. These results will be posted as they become available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT00602667/Prot_SAP_000.pdf